CLINICAL TRIAL: NCT00384579
Title: Pilot Study to Assess the Efficacy of Botulinum Toxin B (Myobloc®) Treatment of Paravertebral Muscles on Pain and Disability in Subjects Suffering From Acute Low Back Pain
Brief Title: Pilot Study to Assess the Efficacy of Botulinum Toxin B on Pain and Disability in Subjects With Acute Low Back Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: No eligible candidates in 2 years of recruiting
Sponsor: United States Department of Defense (U.S. Federal Agency)
Responsible Party: CDR Jack W. Tsao, MD, DPhil, Walter Reed Army Medical Center
Organization: Walter Reed Army Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DCI P05-71031
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-02

CONDITIONS: Low Back Pain
Keywords: back; pain
MeSH Terms: conditions — Low Back Pain; Pain | interventions — rimabotulinumtoxinB

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Botulinum Toxin B
  Interventions: Drug: Botulinum toxin B
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botulinum toxin B — Botulinum Toxin B
  Other Names: Myobloc
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
This study will test the hypothesis that Botulinum toxin B (Myobloc®) treatment reduces pain and disability in subjects suffering from acute low back pain due to an identifiable muscle strain or back trauma occurring 3 to 6 weeks prior to enrollment. The study will also delineate the duration of medication effect and control for any placebo or mechanical trigger-point injection effect by employing a prospective, double-blind, placebo-controlled design.

DETAILED DESCRIPTION:
This study will assess the efficacy of Botulinum Toxin B (Myobloc®) injected into the lumbar paravertebral muscles for reducing pain and disability in subjects suffering from acute low back pain (duration 3 to 6 weeks) arising from an identifiable muscle strain injury or back trauma. The treatment modality and techniques used are based upon three successful prior open-labeled pilot studies done by this research group investigating the effect of Botulinum Toxin A (BOTOX®) on relief of chronic low back pain. This study, however, will employ a prospective, double-blind, randomized, placebo controlled trial to control for any placebo or mechanical trigger-point injection effects. Subjects will also be assessed for 3 months to define the duration of efficacy of Myobloc®. Sixty subjects will be randomly assigned to one of two groups and will then receive either Myobloc® or placebo injection into the lumbar paravertebral muscles. The subjects will be assessed using validated scales for pain and disability prior to injection and weekly to monthly thereafter for three months. All subjects will continue to receive any medication or physiotherapy per standard of care but those treatments will be recorded and controlled for in the data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 to 60 years of age, active duty military, retired military or other DOD beneficiaries eligible for care at military treatment facilities.
* Written informed consent and written authorization for use or release of health and research study information.
* Clear history of an identifiable muscle strain or trauma preceding the onset of low back pain.
* No prior history of vertebral disk disease/condition, sciatica or radiculopathy.
* Normal neurological examination without evidence of radiculopathy.
* Evidence of trigger point tenderness or muscle spasm upon palpation or EMG findings of muscle spasm.
* History of low back pain lasting 3 to 6 weeks from the time of injury or strain.
* VAS score minimum of 5 cm at time of entry into study.
* Ability to follow study instructions and likely to complete all required visits.
* Negative urine pregnancy test prior to the administration of study medication (for females of childbearing potential) (if applicable).

Exclusion Criteria:

* Age less than 18 or greater than 60.
* Not active duty.
* Concomitant use of aminoglycoside antibiotics, curare-like agents, or other agents that might interfere with neuromuscular function.
* Any medical condition that may put the subject at increased risk with exposure to Myobloc®, including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis/motor neuron disease, neuropathy, renal stones, or any other disorder that might interfere with neuromuscular function or produce a similar type of low back pain.
* Females who are pregnant, breast-feeding, or planning a pregnancy during the study, or who think that they may be pregnant at the start of the study, or females of childbearing potential who are unable or unwilling to use a reliable form of contraception during the study.
* Known allergy or sensitivity to any of the components in the study medication.
* Evidence of alcohol or substance abuse in 6 months prior to enrollment.
* Systemic medical conditions (such as thyroid disease, hypertension, bleeding disorders, diabetes, cancers, etc.) that are not currently medically managed or controlled.
* Concurrent participation in another investigational drug or device study or participation in the 30 days immediately prior to study enrollment.
* Any condition or situation that, in the investigator's opinion, may put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study.
* Significant Axis I or II diagnosis determined by a neurologist or psychiatrist in the 6 months prior to entry into the study.
* Duration of low back pain < 3 weeks or > 6 weeks.
* Thoracic or cervical spine pain in the absence of acute low back pain.
* Anesthetic or corticosteroid injection to the lumbosacral spine within 8 weeks of enrollment.
* Spine MRI (any region) positive for acute pathology or evidence of radiculopathy on neurological examination.
* History of back surgery within one year or incomplete resolution of back pain due to a previous injury or surgery.
* Subjects involved in litigation, seeking significant disability for low back pain, or with evident secondary gain as determined by the neurologist through chart review and subject interview.
* Any previous use of Myobloc®, Dysport®, or BOTOX®.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-02; Primary Completion 2010-08 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Significant improvement in lower back pain | 8 weeks

SECONDARY OUTCOMES:
Significant reduction of long term disability | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jack W Tsao, MD, Principal Investigator — Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Wipf JE, Deyo RA. Low back pain. Med Clin North Am. 1995 Mar;79(2):231-46. doi: 10.1016/s0025-7125(16)30065-7. PMID 7877388
- [Background] Frymoyer JW. Predicting disability from low back pain. Clin Orthop Relat Res. 1992 Jun;(279):101-9. PMID 1534720
- [Background] Lew MF, Brashear A, Factor S. The safety and efficacy of botulinum toxin type B in the treatment of patients with cervical dystonia: summary of three controlled clinical trials. Neurology. 2000;55(12 Suppl 5):S29-35. PMID 11188982
- [Background] Rand MJ, Whaler BC. Impairment of sympathetic transmission by botulinum toxin. Nature. 1965 May 8;206(984):588-91. doi: 10.1038/206588a0. No abstract available. PMID 5319286
- [Background] Aoki KR. Review of a proposed mechanism for the antinociceptive action of botulinum toxin type A. Neurotoxicology. 2005 Oct;26(5):785-93. doi: 10.1016/j.neuro.2005.01.017. Epub 2005 Jul 5. PMID 16002144
- [Background] Foster L, Clapp L, Erickson M, Jabbari B. Botulinum toxin A and chronic low back pain: a randomized, double-blind study. Neurology. 2001 May 22;56(10):1290-3. doi: 10.1212/wnl.56.10.1290. PMID 11376175
- [Background] Aoki KR. Pharmacology and immunology of botulinum toxin serotypes. J Neurol. 2001 Apr;248 Suppl 1:3-10. doi: 10.1007/pl00007816. PMID 11357237